CLINICAL TRIAL: NCT06191900
Title: Single Arm Clinical Study of Autologous Tumor Infiltrating Lymphocyte Injection (GT201) in the Treatment of Advanced Gynecological Tumors (advanced Cervical Cancer)
Brief Title: Clinical Study of GT201 in the Treatment of Advanced Gynecological Tumors (advanced Cervical Cancer)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-201-001
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Adult; Gynecological Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT201 treatment group (Experimental)
  Interventions: Biological: Autologous tumor infiltrating lymphocyte injection（GT201）

INTERVENTIONS:
Biological: Autologous tumor infiltrating lymphocyte injection（GT201） — GT201 treatment for advanced gynecological tumors (advanced cervical cancer)

SUMMARY:
This study is an early exploration clinical study with one arm.

The study consists of two stages, namely the dose escalation stage and the dose extension stage:

ELIGIBILITY:
Inclusion Criteria:

* 1. The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), must have the ability to understand the requirements of the study;
* 2.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies. The separated tissues mass weighing ≥1.0g (either of single lesion origin or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible;

Exclusion Criteria:

* 1.The patient who has any active autoimmune disease, history of autoimmune disease, need for systemic steroid hormones or a condition requiring immunosuppressive drug therapy (>10 mg/day of prednisone or equivalent hormone);
* 2. Arterial/venous thrombotic events within 3 months prior to enrollment, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 3.Active infections requiring treatment with systemic anti-infectives (except for topical antibiotics); or those with unexplained fever > 38.5℃ occurring during the screening period, except for tumor fever;
* 4. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 5.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adcersed events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection（GT201) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adcersed events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No